CLINICAL TRIAL: NCT02380053
Title: Proof of Concept Study to Assess the Differential Effects of Chronic Beta-blockade (Celiprolol Versus Bisoprolol) on Cardiopulmonary Outcomes at Rest and During Exercise in Chronic Obstructive Pulmonary Disease
Brief Title: Chronic Beta-blockade and Cardiopulmonary Exercise in COPD
Acronym: CPET1
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Dundee (Other)
Responsible Party: Principal Investigator, William J Anderson, Consultant Respiratory Physician and Honorary Senior Lecturer, University of Dundee
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CPET1; 2015-000207-13 (EudraCT Number); 2012RC22 (Other: Sponsor (NHS Tayside/University of Dundee))
Record Dates: First submitted 2015-02-19; First posted 2015-03-05 (Estimated); Last update posted 2019-06-24 (Actual); Status verified 2019-06

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Beta-blocker; Cardiopulmonary exercise testing
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Bisoprolol; Celiprolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bisoprolol (Experimental): 2.5mg once daily for 2 weeks then 5mg once daily for 2 weeks.
  Interventions: Drug: Bisoprolol
- Celiprolol (Experimental): 200mg once daily for 2 weeks then 400mg once daily for 2 weeks.
  Interventions: Drug: Celiprolol

INTERVENTIONS:
Drug: Bisoprolol — 2 weeks of Bisoprolol 2.5mg daily then 2 weeks Bisoprolol 5mg daily
  Arms: Bisoprolol
Drug: Celiprolol — 2 weeks of Celiprolol 200mg daily then 2 weeks Celiprolol 400mg daily
  Arms: Celiprolol

SUMMARY:
What are the differential effects of beta-blockers on lung and heart function during exercise in chronic obstructive pulmonary disease (COPD)? COPD is a major cause of illness and death. Not only do these individuals suffer from lung disease, but COPD often leads to other illnesses, particularly heart disease. Beta-blockers very successfully treat heart disease. It is therefore logical that one would want to use this treatment in COPD patients with heart disease too. However, there has always been concern that beta-blockers could cause significant problems in COPD by worsening lung function, as these can have the opposite effect to inhalers used to treat COPD that open up airways. Pointedly, there is increasing evidence that despite this problem, COPD patients who have been prescribed beta-blockers have been shown to gain benefit particularly in terms of preventing death.

In this study, the investigators therefore want to examine which beta-blocker might be the safest for COPD patients, as each work slightly differently. Some beta-blockers may have a more beneficial effect on airways than others, whilst still benefitting the heart. The investigators will study two different beta-blockers; one that potentially narrows airways and one that potentially opens airways. The investigators will be using cardiopulmonary exercise testing (an exercise bike that measures both heart and lung function during exercise) to look for differences between both beta-blockers primarily in terms of lung function but also with information about the heart. The investigators will recruit people with moderate to severe COPD who are able to complete a cycle exercise test through their respiratory research department. The study will last for 10-12 weeks with 5 main visits to the department for serial exercise tests, breathing tests, simple heart function tests and simple blood tests that will tell the investigators what other effects these beta-blockers are having on the heart and lungs.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is a major cause of illness and death. In fact, by 2020, the World Health Organization predicts that COPD will become the third leading cause of death (currently fourth), and the fifth leading cause of disability (currently twelfth) worldwide. COPD and cardiovascular (heart) disease are intertwined due to the associated risk of smoking related atherosclerosis. Beta-blockers are generally avoided in COPD patients due to the associated risk of worsening lung function and acute bronchospasm (airway narrowing) due to beta-2-receptor blockade. Despite these concerns a recent Cochrane review has shown that chronic beta-blockade with "cardioselective" beta-blockers (for example bisoprolol) that preferentially block beta-1 (mostly heart) over beta-2 (mostly airway) receptors are well tolerated with less beta-2-blockade and subsequently less bronchospasm.

Furthermore, observational studies evaluating the impact of beta-blocker use in COPD patients have shown benefits on survival with beta-blockers. We have published retrospective data from 5,977 patients with COPD with a mean follow up of 4.35 years, showing that patients using beta-blockers (88% cardio-selective) produced a 22% overall reduction in death as well as significant reductions in respiratory hospital admissions and oral steroid use.

Beta-blockers are pharmacologically different and there now needs to be an assessment of the clinical consequences of different beta-blockers in COPD. Despite being "cardioselective", bisoprolol still shows significant beta-2-receptor blockade at usual treatment doses, which results in a significant worsening in Forced Expiratory Volume in 1second - FEV1 (a major marker of lung function) following chronic use. Celiprolol however is a unique beta-blocker which in addition to its beta-1-receptor blockade has partial beta-2-agonist activity and therefore it does not cause bronchoconstriction or interact with short and long acting beta-agonist inhalers which are the mainstay of COPD treatment. Thus celiprolol might confer an ideal profile for use in COPD (i.e. good for heart and not detrimental to lungs), especially in more severe patients where even a small fall in FEV1 might have significant consequences on their breathing and exercise capacity.

Poor exercise tolerance is associated with worsening quality of life and increased risk of death and thus provides a valuable surrogate marker of death. Worsening respiratory symptoms in COPD patients are more commonly seen on exertion than at rest, and associated with abnormal increases in lung volumes where air that is breathed in becomes trapped and cannot completely escape when breathing out (dynamic hyperinflation).

Cardiopulmonary exercise testing provides a global assessment of both respiratory (lung) and cardiovascular (heart) response to exercise. Whilst studies have shown a worsening of dynamic hyperinflation with bisoprolol, due to their differing pharmacological properties it might be that celiprolol will not result in worsening dynamic hyperinflation, whilst also demonstrating improvement in cardiovascular outcomes such as stroke volume (the pump function of the heart) and heart rate recovery following exercise. Whether these effects result in an improved exercise tolerance is unknown. Another interesting property of celiprolol is reduced cholesterol and increased High Density Lipoprotein (HDL) fraction conferred by partial beta-2-agonist activity. We will also measure serum markers of cardiac dysfunction (B-type Natriuretic Peptide (BNP) and Galectin-3) and their response to beta-blockade which to the investigators' knowledge has never been performed in a COPD study.

With regards to measuring cardiovascular outcomes of cardiac output and stroke volume, the investigators plan to use a novel non-invasive monitor which is based on the phenomenon of bioreactance that occurs when a small alternating current is passed through the chest. To the investigators' knowledge this device has never been used when assessing cardiovascular response to beta-blockers during exercise, but it is safe and easy to perform at the same time as the standard exercise test.

The investigators therefore wish to assess the relative effects of both celiprolol and bisoprolol in COPD patients and establish whether the proposed benefits on survival with beta-blockers in COPD are reflected in improved cardiovascular and respiratory response to exercise and importantly exercise tolerance. The investigators also want to see if celiprolol is superior to bisoprolol on these markers (particularly lung function) as described above.

The information gathered from this study will be invaluable as it will provide further information about the effects of beta-blockers in COPD and will be used to pump-prime larger long-term studies examining the effects of beta-blockers on survival in many more COPD patients.

Hypothesis The null hypothesis is that there is no difference between bisoprolol and celiprolol in terms of cardiorespiratory outcomes during incremental exercise testing in patients with moderate to severe COPD - specifically no difference in the proposed primary outcome measure of dynamic hyperinflation during cycle endurance testing.

Design The investigators have chosen a randomised crossover design to answer this question because it is unknown which, if either, beta-blocker might be better for lung function and exercise capacity in moderate to severe COPD patients. The crossover design allows the use of the same patients as their own comparators, thus allowing the investigators to expose fewer patients to these medications with the same statistical power as a parallel group study (different patients in each group). Each participant will therefore receive both treatments in sequence but with their initial one decided at random using a randomisation algorithm. Importantly the investigators have not used a placebo control arm here, as it is already known that beta-blockers are of benefit to COPD patients (particularly those with cardiovascular disease) whereas placebo provides no benefit. In other words the investigators are drilling down to see which particular medication has the most beneficial therapeutic profile. The justification for using open-label beta-blockers is that this is a pilot study and it helps to keep the overall costs of the study down at this stage of investigation.

Methods The investigators will perform a randomised, cross-over, open label trial of bisoprolol versus celiprolol with 10 people who have moderate to severe COPD. The study will last between 10-12 weeks for each person. Potential participants will be recruited from our existing database of volunteers with COPD, contacted either by telephone, email or post and invited to participate. Those invited will receive a written patient information document detailing the requirements of the study and the extent of their participation before attending for a screening visit. Participants will be given at least 24hours to read the information document before deciding whether or not they agree to be screened. The study will include 5 visits to the department (including the screening visit) for the various tests outlined below. Each visit may last for around 3 hours. If participants agree to coming along for a screening visit, they will be asked to withhold any long-acting bronchodilators for 48hours and short acting bronchodilators for 6 hours as is standard practice when confirming the diagnosis of airway obstruction / COPD using clinical pulmonary function measurements.

Screening Visit At the screening visit, the information document will be discussed with the participant and written informed consent will be obtained if they agree to take part in the study. The following will then be performed: a general medical examination by a doctor; a pregnancy test for all females; lung function measurements (spirometry, impulse oscillometry, reversibility to salbutamol); heart function measurements (resting ECG [electrocardiogram], echocardiogram where possible if not done in last year); vital signs (oxygen levels, blood pressure, pulse); 'practice' cardiopulmonary exercise test (to confirm ability to cycle and to counter any 'learning effect' from future baseline exercise test); baseline blood tests. Inhaler technique will also be assessed and confirmed adequate. Participants found to be eligible for the remainder of the study after these tests will proceed through a 1 week run-in period on their usual medications before coming back for the first (baseline) visit. Those who do not fulfil the study criteria will continue on their usual medication and their General Practitioner (GP) informed of any medically relevant data. Eligible participants will be provided with portable monitors to measure their own lung function, pulse and oxygen saturations at home twice daily to be recorded in a daily diary which will also include details of their reliever use and symptoms. This diary will be kept throughout the study.

Study visits Prior to participants attending for their first (baseline) study visit they will be asked to only withhold their short-acting reliever inhaler for 6 hours. Participants will not be required to withhold any long-acting bronchodilators for study visits as we are assessing any effects of the beta-blockers in addition to these standard treatments and we will have confirmed the diagnosis of COPD at the screening visit. Diary cards will be reviewed and the following measurements will be recorded at visit 1: resting lung function (impulse oscillometry, spirometry, whole body plethysmography); resting ECG; vital signs; St George's Respiratory Questionnaire (disease specific quality of life questionnaire); blood sample (BNP, Galectin, Cholesterol/HDL, Creatine Kinase (CK), Potassium); cardiopulmonary exercise test. Provided the participant's measurements still correspond to the inclusion and exclusion criteria for the study, they will be randomised to one of the two beta-blocker treatments: Bisoprolol (2.5mg daily for 2 weeks, then 5mg daily for approximately 2 weeks) OR Celiprolol (200mg daily for 2 weeks, then 400mg daily for approximately 2 weeks). Beta-blockers will be up-titrated at home after 2 weeks with advice about contacting us if side effects develop. Participants will be contacted both before and after this up titration either by telephone or email. However, if adverse effects occur on the higher dose, then participants will be allowed to drop back to the lower dose for the remainder of the study period. At the end of each treatment period, study measures will be repeated as above. After visit 2 participants will have an approximately 1 week washout period prior to being given the alternate beta-blocker treatment.

End of study After visit 4 each participant will have completed the study and they will be returned to their usual medications. The overall study will be complete when the last enrolled participant completes the protocol.

Analysis and final reporting All analyses will be performed at the end of the study. There will be no interim analysis. The report will be published in a high impact peer reviewed journal.

ELIGIBILITY:
Inclusion Criteria:

* Male and female volunteers aged 40-80 years
* Stable moderate to severe COPD (Global initiative on Obstructive Lung Disease [GOLD] stage 2/3)
* Post-bronchodilator FEV1 30-80% predicted
* FEV1/FVC ratio <70%
* Stable defined as no exacerbation in previous 1 month
* Smoking history ≥10 pack-years
* Oxygen saturations ≥92% on room air at rest
* Electrocardiogram demonstrating sinus rhythm.

Exclusion Criteria:

* Use of domiciliary oxygen
* History of other primary obstructive lung disease including asthma or bronchiectasis
* Hospitalisation with exacerbation of COPD within past 3 months
* History of unstable angina, uncontrolled hypertension or heart failure (New York Heart Association class 3-4)
* Overt clinical signs of right heart failure
* Average resting systolic BP<110mmHg or average resting HR<55bpm
* Pregnancy or lactation
* Known or suspected sensitivity to/intolerance of investigational medicinal product
* Inability to comply with compulsory aspects of protocol
* Any degree (first, second or third) of heart block
* Sino-atrial block
* Sick sinus syndrome
* Severe forms of peripheral arterial occlusive disease or severe forms of Raynaud's syndrome
* Untreated phaeochromocytoma
* Severe renal impairment (eGFR<15ml/min)
* Concomitant prescription of beta-blockers, rate-limiting calcium channel blockers, digoxin, amiodarone
* Any clinically significant medical condition that may endanger the health or safety of the participant, or jeopardise the protocol
* Participation in another trial within the previous 30 days

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2016-06-07 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Change in Inspiratory Capacity (IC) from rest to isotime peak. | Baseline to 4 weeks
  The primary outcome for this study will be the difference from baseline in the change in Inspiratory Capacity (IC) from rest to isotime peak (i.e. same time point during endurance exercise test) between beta-blocker treatments at 4 weeks. This will evaluate any differences in dynamic hyperinflation during exercise between treatments.

SECONDARY OUTCOMES:
Exercise outcome: Oxygen uptake at peak exercise (VO2peak) | Baseline to 4 weeks.
Exercise outcome: Anaerobic threshold (AT) | Baseline to 4 weeks.
Exercise outcome: Heart rate | Baseline to 4 weeks.
Exercise outcome: Heart rate reserve (HRR) | Baseline to 4 weeks.
Exercise outcome: Heart rate recovery (HRrec) | Baseline to 4 weeks.
Exercise outcome: Respiratory rate | Baseline to 4 weeks.
Exercise outcome: Breathing reserve | Baseline to 4 weeks.
Exercise outcome: Ventilatory equivalent for oxygen at anaerobic threshold | Baseline to 4 weeks.
  Measure of ventilatory efficiency
Exercise outcome: Ventilatory equivalent for carbon dioxide at anaerobic threshold | Baseline to 4 weeks.
  Measure of ventilatory efficiency
Exercise outcome: Pulse oximetry at peak exercise | Baseline to 4 weeks.
Exercise outcome: Oxygen pulse (O2P) | Baseline to 4 weeks.
  Surrogate for stroke volume
Exercise outcome: Total exercise time | Baseline to 4 weeks.
Non-invasive cardiac output measure: Stroke volume | Baseline to 4 weeks
Non-invasive cardiac output measure: Cardiac output | Baseline to 4 weeks
Non-invasive cardiac output measure: Cardiac Index | Baseline to 4 weeks
Spirometry: Forced expiratory volume in 1s (FEV1) | Baseline to 4 weeks
  Spirometry, Impulse oscillometry, whole body plethysmography
Spirometry: Forced Vital Capacity (FVC) | Baseline to 4 weeks
Spirometry: Forced expiratory flow between 25-75% of FVC | Baseline to 4 weeks
Spirometry: FEV1/FVC ratio | Baseline to 4 weeks
Impulse oscillometry: Resistance at 5 Hertz (R5) | Baseline to 4 weeks
  Measure of total airway resistance
Impulse oscillometry: Resistance at 20 Hertz (R20) | Baseline to 4 weeks
  Measure of large airway resistance
Impulse oscillometry: Reactance at 5 Hertz (X5) | Baseline to 4 weeks
  Measure of airway compliance
Impulse oscillometry: Area under the curve | Baseline to 4 weeks
  Measure of small airways resistance
Impulse oscillometry: Frequency of resonance | Baseline to 4 weeks
  Measure of small airways resistance
Whole body plethysmography: Total lung capacity | Baseline to 4 weeks
Whole body plethysmography: Residual volume | Baseline to 4 weeks
  Measure of air trapping in the lungs
Supine blood pressure | Baseline to 4 weeks
Erect blood pressure | Baseline to 4 weeks
Change in blood B-natriuretic peptide levels | Baseline to 4 weeks
Change in blood Galectin levels | Baseline to 4 weeks
Change in blood Cholesterol/HDL levels | Baseline to 4 weeks
Change in blood creatine kinase levels | Baseline to 4 weeks
Change in blood potassium levels | Baseline to 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: William J Anderson, MBCHB, Principal Investigator — University of Dundee / NHS Tayside
Locations (1):
- Asthma and Allergy Research Group, Ninewells Hospital and Medical School, University of Dundee, Dundee, United Kingdom

REFERENCES:
- [Derived] Anderson W, Short P, Ross R, Lipworth BJ. Bisoprolol versus celiprolol on dynamic hyperinflation, cardiopulmonary exercise and domiciliary safety in COPD: a single-centre, randomised, crossover study. BMJ Open Respir Res. 2023 Jul;10(1):e001670. doi: 10.1136/bmjresp-2023-001670. PMID 37451701